CLINICAL TRIAL: NCT05851950
Title: RUFUS - a Randomized Mixed Methods Pilot Clinical Trial Investigating the Relevance and Feasibility of Rumination-focused Cognitive Behavioral Therapy in the Treatment of Patients With Emergent Psychosis Spectrum Disorder
Brief Title: RUFUS - Group Rumination-focused CBT for Negative Symptoms
Acronym: RUFUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 05851950
Record Dates: First submitted 2023-05-01; First posted 2023-05-10 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Psychotic Disorders
MeSH Terms: conditions — Psychotic Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rumination-focused cognitive behavioural group therapy (Experimental): 1 individual in-take session, 11 sessions of rumination-focused cognitive behavioural group therapy, 1 individual closing session.
  Interventions: Other: group rumination focused cognitive behavioural therapy
- Treatment as usual (Active Comparator): standard OPUS treatment. OPUS treatment is handled by an interdisciplinary OPUS team and consists primarily of medical treatment, psychoeducation, training in symptom management and social skills as well as family discussions. All patients in OPUS have a contact doctor and a contact person who is responsible for coordinating the treatment and collaborating with municipal bodies.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Other: group rumination focused cognitive behavioural therapy — Psychotherapy
  Arms: rumination-focused cognitive behavioural group therapy
Other: Treatment as usual — opus treatment
  Arms: Treatment as usual

SUMMARY:
Abstract - --

Introduction:

Psychosis spectrum disorders are characterized by both positive and negative symptoms, but whereas there is good effect of treatment on positive symptoms, there is still a scarcity of effective interventions aimed at reducing negative symptoms. Rumination has been proposed as an important and fundamental factor in the development and maintenance of symptoms across psychiatric diagnoses, and there is a need to develop effective interventions targeting rumination behaviors and negative symptoms in patients with psychotic disorders. The aim of the current study is to investigate the feasibility and acceptability of group rumination-focused cognitive behavioral therapy (RFCBT) in the treatment of young people with psychosis spectrum disorders as well as investigating potential indications of treatment efficacy.

Methods and analysis: The study is a mixed-method clinical randomized controlled pilot trial with a target sample of 60 patients, who are randomized to either receive 13 weeks of group CFCBT or 13 weeks of treatment as usual (TAU). All patients are examined at the start of the project and at the 13-week follow-up. The researcher will compare changes in outcomes from baseline to posttreatment between group CFCBT and TAU. In addition, qualitative analyzes are carried out to explore feasibility and acceptability and to uncover the patients' experience of receiving the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with a psychosis spectrum disorder (ICD-10 F2x)
2. At least 8 months left of their OPUS treatment
3. The presence of rumination behavior as assessed by a score of minimum 30 on the Perseverative Thinking Questionnaire (PTQ)
4. Danish-speaking

Exclusion Criteria:

1. Substance abuse or positive symptoms that make participation in therapy difficult
2. Severe suicidal thoughts/behavior
3. Lacks capacity to consent
4. Mild, moderate, or severe intellectual disability (IQ ˂ 70)
5. Planned adjustment of antidepressant and/or antipsychotic treatment (noted in the patient's medical record)

Ages: 18 Years to 37 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
the Brief Negative Symptoms Scale (BNSS) | up to 20 weeks
  Assessment of negative symptoms on a scale from 0-78

SECONDARY OUTCOMES:
Perseverative Thinking Questionnaire (PTQ) | up to 20 weeks
  Measuring frequency of rumination. Resulting in a total score of 0-60.
Ruminative Response Scale (RRS) | up to 20 weeks
  Measuring levels of rumination in relation to depression. Resulting in a total score of 22-88.
Social Functioning Scale (SFS) | up to 20 weeks
  Measuring level of functioning on a scale from of 0-228
Scale for the assessment of positive symptoms (SAPS) | up to 20 weeks
  Measuring presence of positive symptoms on a scale from 0-170
Calgary depression scale (CDS) | up to 20 weeks
  Measuring depressive symptoms on a scale from 0-27
Behavior Rating Inventory of Executive Function (BRIEF) | up to 20 weeks
  Measuring executive functioning on a scale from 75-225

CONTACTS AND LOCATIONS:
Overall Officials: Louise B Glenthøj, Principal Investigator — Mental health center of Copenhagen
Locations (1):
- Mental Health Centre Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No